CLINICAL TRIAL: NCT05111171
Title: The Guiding Value of Ultrasound and Radial Arteriography in the Selection of Sheath Size for Transradial Coronary Intervention: A Single-center Clinical Study
Brief Title: The Guiding Value of Ultrasound and Radial Arteriography in the Selection of Sheath Size for Transradial Coronary Intervention
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Chief leader of CCU, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 017
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Condoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6F sheath CAG group: No PCI is required, only diagnostic CAG is required.
  Interventions: Device: sheath
- 6F sheath PCI group: PCI is required, simple lesions are group.
  Interventions: Device: sheath
- 7F sheath PCI group: PCI is required for the complicated disease.
  Interventions: Device: sheath

INTERVENTIONS:
Device: sheath — Senior interventional doctors interpret the CAG results and group according to their clinical experience: (1) No PCI is required, only diagnostic CAG is required, which is group ①6F sheath CAG group; (2) PCI is required, simple lesions are group ②6F sheath PCI group, the 6F sheath is still used for PCI; (3) PCI is required for the complicated disease and use 7F sheath, as the 7F sheath PCI group is the group ③, and the 7F sheath is replaced for PCI.

SUMMARY:
Coronary angiography is a relatively safe and reliable invasive diagnostic technique, clinically considered the "gold standard" for diagnosing coronary heart disease. In 1989, Canadian doctor Campeau performed trans-radial angiography (TRA) for the first time percutaneous puncture of the radial artery. In 1993, Dutch doctor Keimeneij and others completed the first trans-radial coronary intervention (trans-radial intervention, TRI) . After nearly 30 years of clinical practice, the radial artery approach has become the first choice for coronary intervention and treatment. Compared with the femoral artery approach, the radial artery approach has the advantages of fewer traumas, less risk of bleeding, shorter hospital stay, and patients' early mobility. However, there are also few disadvantages of the radial access, such as small inner diameter, repeated puncture prone to spasm, limiting the implantation of larger sheaths to treat complex coronary artery diseases and postoperative complications such as thickening and stenosis and occlusion of the radial artery. The incidence is higher, and so on.Previous studies have found that the mismatch between the radial artery's inner diameter and the sheath's diameter is an essential factor that causes complications such as thickening, stenosis, and occlusion of the radial artery after intervention. Patients with coronary heart disease often need to repeat coronary interventional examinations and treatments. To ensure the radial artery route and avoid complications such as radial artery occlusion (RAO) after intervention for repeated use. It is worthy of attention. At present, in clinical ascending coronary angiography (CAG) or coronary interventional therapy (PCI), most of the radial artery sheath sizes are not selected according to the diameter of the patient's radial artery. The surgeon is only subjectively based on the patient's radial artery pulsation strength and coronary artery pulsation. It depends on the complexity of the pulse pathology. The incidence of radial artery occlusion reported in previous studies is 5%-38%. Most of these studies only rely on clinical forearm examination and pulse palpation without vascular ultrasound, radial angiography, and other imaging examinations to assess catheter placement. The degree of patency of the posterior radial artery has caused considerable differences in the reported incidence of radial artery occlusion. However, PCI treatment of complex lesions such as bifurcation, high calcification, severe distortion, chronic total occlusion, etc., usually requires a 7F sheath to provide better support and convenient equipment delivery. Still, the latter has the following problems: on the one hand, patients' pain, vasospasm, and other reasons can easily lead to failure of the radial artery sheath grafting; on the other hand, although the 7F sheath is used to complete PCI for complex lesions, the postoperative Radial artery occlusion is prone to occur, resulting in long-term failure to undergo re-radial artery angiography or PCI treatment.The innovation of this study lies in the use of ultrasound and radial angiography for the measurement of the inner diameter of the patient's radial artery, to examine the distribution of the inner diameter of the radial artery, and to predict the cut-off value of the radial artery inner diameter for successful sheath implantation and the inner diameter resection of the radial artery occlusion after the operation. The point value provides an evidence-based basis for selecting the sheath size of the radial artery in the future to achieve the clinical purpose of protecting the radial artery for repeated use.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are diagnosed or suspected of having coronary heart disease;
2. Patients undergoing first time selective interventional surgery via the right radial artery;
3. Those who can understand the purpose of this experiment, participate in this study voluntarily, and sign an informed consent form.

Exclusion Criteria:

1. Have a history of PCI through the right radial artery;
2. Those with deformity, trauma, or amputation of the right upper limb;
3. Those who have negative Allen's test;
4. There are other contraindications to coronary angiography surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study adopts a continuous enrollment method. It is estimated that 500 patients will be enrolled within the study period.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The cut-off value of the radial artery inner diameter, successfully implanted with 6F and 7F sheath. | 30days
The cut-off value of the radial artery diameter, at which the radial artery occlusion occurred in the 6F and 7F sheath groups. | 30days

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campeau L. Percutaneous radial artery approach for coronary angiography. Cathet Cardiovasc Diagn. 1989 Jan;16(1):3-7. doi: 10.1002/ccd.1810160103. PMID 2912567
- [Result] Kiemeneij F, Laarman GJ. Transradial artery Palmaz-Schatz coronary stent implantation: results of a single-center feasibility study. Am Heart J. 1995 Jul;130(1):14-21. doi: 10.1016/0002-8703(95)90229-5. PMID 7611104
- [Result] Rao SV, Cohen MG, Kandzari DE, Bertrand OF, Gilchrist IC. The transradial approach to percutaneous coronary intervention: historical perspective, current concepts, and future directions. J Am Coll Cardiol. 2010 May 18;55(20):2187-95. doi: 10.1016/j.jacc.2010.01.039. PMID 20466199
- [Result] Kanei Y, Kwan T, Nakra NC, Liou M, Huang Y, Vales LL, Fox JT, Chen JP, Saito S. Transradial cardiac catheterization: a review of access site complications. Catheter Cardiovasc Interv. 2011 Nov 15;78(6):840-6. doi: 10.1002/ccd.22978. Epub 2011 May 12. PMID 21567879
- [Result] Pancholy S, Coppola J, Patel T, Roke-Thomas M. Prevention of radial artery occlusion-patent hemostasis evaluation trial (PROPHET study): a randomized comparison of traditional versus patency documented hemostasis after transradial catheterization. Catheter Cardiovasc Interv. 2008 Sep 1;72(3):335-340. doi: 10.1002/ccd.21639. PMID 18726956
- [Result] Stella PR, Kiemeneij F, Laarman GJ, Odekerken D, Slagboom T, van der Wieken R. Incidence and outcome of radial artery occlusion following transradial artery coronary angioplasty. Cathet Cardiovasc Diagn. 1997 Feb;40(2):156-8. doi: 10.1002/(sici)1097-0304(199702)40:23.0.co;2-a. PMID 9047055
- [Result] Sanmartin M, Gomez M, Rumoroso JR, Sadaba M, Martinez M, Baz JA, Iniguez A. Interruption of blood flow during compression and radial artery occlusion after transradial catheterization. Catheter Cardiovasc Interv. 2007 Aug 1;70(2):185-9. doi: 10.1002/ccd.21058. PMID 17203470
- [Result] Cubero JM, Lombardo J, Pedrosa C, Diaz-Bejarano D, Sanchez B, Fernandez V, Gomez C, Vazquez R, Molano FJ, Pastor LF. Radial compression guided by mean artery pressure versus standard compression with a pneumatic device (RACOMAP). Catheter Cardiovasc Interv. 2009 Mar 1;73(4):467-72. doi: 10.1002/ccd.21900. PMID 19229978
- [Result] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409
- [Result] Yan ZX, Zhou YJ, Zhao YX, Zhou ZM, Yang SW, Wang ZJ. Anatomical study of forearm arteries with ultrasound for percutaneous coronary procedures. Circ J. 2010 Apr;74(4):686-92. doi: 10.1253/circj.cj-09-0577. Epub 2010 Mar 3. PMID 20197630
- [Result] Uhlemann M, Mobius-Winkler S, Mende M, Eitel I, Fuernau G, Sandri M, Adams V, Thiele H, Linke A, Schuler G, Gielen S. The Leipzig prospective vascular ultrasound registry in radial artery catheterization: impact of sheath size on vascular complications. JACC Cardiovasc Interv. 2012 Jan;5(1):36-43. doi: 10.1016/j.jcin.2011.08.011. PMID 22230148